CLINICAL TRIAL: NCT05313113
Title: The Effect of Self-made Fetal Movement and Position Tracking on Prenatal Attachment and Pregnancy Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, AYSUN BADEM, Assistant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KKYFHTPBVGDE85
Record Dates: First submitted 2022-02-07; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Prenatal Attachment; Fetal Position Tracking; Distress
Keywords: Prenatal attachment; Pregnancy; Fetal Position Tracking; Fetal Movement Count; Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the first stage, pregnant women were trained to implement fetal movement count and position tracking. The training was provided face to face and lasted 30-45 minutes. How to determine the position of the fetus and I. and II. Leopold maneuvers are also taught. In the second stage, the pregnant women were interviewed twice a week by telephone.Thus, it was provided that pregnant women had fetal tracked at least once a day, at any time of the day, when the fetus was awake and most active, in a suitable position and a comfortable environment, for at least 15-20 minutes continuously for four weeks. Pregnant women phoned the researcher when they wanted. At the same time, the participants continued to their routine prenatal care.
  Interventions: Behavioral: Experimental
- Control Group (No Intervention): The pregnant women continued to their routine prenatal care. No intervention was applied to the pregnant women in addition to their routine prenatal care.The pregnant women were called about whether continuing their routine care or having any problems during the research.

INTERVENTIONS:
Behavioral: Experimental — Pregnant women were trained to implement fetal movement count and position tracking. The training was provided face to face and lasted 30-45 minutes. The training content included topics such as setting a comfortable environment and suitable position for the pregnant, when the fetus is active and asleep during the day, how to count and how to evaluate the movements. How to determine the position of the fetus and I. and II. Leopold maneuvers are also taught. In the second stage, the pregnant women were interviewed twice a week by telephone.Thus, it was provided that pregnant women had fetal tracked at least once a day, at any time of the day, when the fetus was awake and most active, in a suitable position and a comfortable environment, for at least 15-20 minutes continuously for four weeks. Pregnant women phoned the researcher when they wanted. At the same time, the participants continued to their routine prenatal care.
  Arms: Experimental group

SUMMARY:
This study was conducted to determine the effect of self-made fetal movement counting and fetal position tracking on prenatal attachment and prenatal distress.

DETAILED DESCRIPTION:
Attachment, which is the basis for establishing social relationships, is the intense feelings that people develop towards the people they consider important. These strong emotions begin with the mother, who is the first person to interact with the individual. When the woman learns that she is pregnant, she becomes curious about her baby, dreams related to the baby, and starts communicating with her baby. Therefore, when baby movements are felt, prenatal attachment becomes stronger, and the cornerstones of attachment are formed.

The early development of safe and positive attachment composes the basis of healthy development. In the later years of childhood, safe attachment is effective on healthy processes, such as being more positive, establishing close, constructive and respectful relationships, and a high sense of trust, while unsafe attachment is associated with emotional, social, physical, and mental psychopathologies.

The mother's touching her baby over her abdomen, trying to guess the parts of the baby, following baby movements, communicating with the baby by focusing and spending private time with the baby increase the physical and psychological contact with the baby. Thus, the baby can be accepted by the mother as an individual, and the attachment between the mother and baby can increase.

Fetal movement counting is defined as tracking uninterrupted fetal movements for at least 15-20 minutes by lying on the left side in a calm environment at any time during the day when this baby is awake. Fetal position tracking is described as trying to guess the parts of the baby by placing the mother's hand on the abdomen. Thanks to fetal movement and position tracking, the state of fetal health can be determined, mother-baby attachment can be increased, and pregnancy distress can be reduced. Pregnant women also may experience negative emotions because of stress, anxiety, anxious anticipation, deterioration of body perception, adaptation to the new situation, anxiety about being a parent, increasing financial needs, fear of birth, and insufficient social support. Hence pregnancy distress can prevent a pleasant pregnancy period and can cause a negative effect on mother-baby attachment.

In order to increase attachment, mothers can be trained on fetal movement and position tracking. This training can be integrated into routine prenatal care since it can be taught quickly. Moreover, it is helpful and economically viable and providing early recognition of fetal risk.

This study was conducted to determine the effect of self-made fetal movement and position tracking on prenatal attachment and pregnancy distress.

ELIGIBILITY:
Inclusion Criteria:

* least literate
* between the ages of 19-35
* Effective communication
* first pregnancy
* having a single fetus
* Pregnancy week between 24 and 28.

Exclusion Criteria:

* Pregnancy using assisted reproductive techniques
* Having a risky pregnancy (preeclampsia, placenta previa, gestational diabetes etc.)
* Pregnant women with a chronic disease (heart, systemic, circulatory disorder, psychiatric, etc.) were not included in the study.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — focused on pregnancy women
Enrollment: 85 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
The mean prenatal attachment level (mean±SD) | between 24-28 gestational weeks and after 30 days
  The mean prenatal attachment was assessed using ''Prenatal attachment inventory''. The inventory consists of 21 Likert-type items. Each item is scored between 1 and 4. Therefore, the minimum score of the inventory is 21, while the maximum score of the inventory is 84. The pregnant between 24-28 gestational weeks were filled with face-to-face interviews at the first interview and 30 days after the training.
The mean pregnancy distress level (mean±SD) | between 24-28 gestational weeks and after 30 days
  The mean pregnancy distress was assessed using "Pregnancy Distress Scale".The TPDS consists of 16 items and two sub-dimensions as negative affect and partner involvement. The TPDS is 4-point likert type. Each item is scored between 0 and 3. Thus, the total score of TPDS is ranged between 0 and 48 on the scale. The higher the score, the higher the pregnancy distress. The pregnant between 24-28 gestational weeks were filled with face-to-face interviews at the first interview and 30 days after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badem A, Mucuk S. The effect of self-evaluation of foetal movement and position tracking on prenatal attachment and distress. J Reprod Infant Psychol. 2024 Jun;42(3):439-448. doi: 10.1080/02646838.2022.2117290. Epub 2022 Sep 1. PMID 36047609